CLINICAL TRIAL: NCT01286727
Title: Multicenter Pilot Study of BB3 to Improve Renal Function in Patients With Signs and Symptoms of Significant Renal Injury After Kidney Transplantation and at Risk for Dialysis
Brief Title: Study to Improve Renal Function After Kidney Transplantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Angion Biomedica Corp (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 001-09; 2R44DK066654 (NIH)
Record Dates: First submitted 2011-01-27; First posted 2011-01-31 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2014-10

CONDITIONS: Delayed Graft Function
MeSH Terms: conditions — Delayed Graft Function

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal Saline (Placebo Comparator): Placebo
- BB3 (Active Comparator)
  Interventions: Drug: BB3

INTERVENTIONS:
Drug: BB3 — intravenous drug
  Arms: BB3

SUMMARY:
The objective of the study is to evaluate the safety and activity of a investigational drug in improving renal function in patients who have undergone renal transplantation and have signs and symptoms of significant renal injury and are at risk for dialysis.

DETAILED DESCRIPTION:
Delayed graft function (DGF) is generally defined as the need for dialysis during the first 7 days after transplantation although the definition can also include failure to improve preexisting renal function. DGF is an important problem in renal allograft transplantation that affects approximately 25% of transplanted cadaveric kidneys. It has generally been observed that delayed graft function has been associated with reduced graft survival. In addition to an association of DGF with graft loss, DGF imposes an economic burden due to prolonged hospitalization and dialysis. The strongest association with occurrence of DGF is ischemia around the time of transplantation. Aside from approaches to minimize ischemia time and use of antibody induction, there are no good specific therapeutic options to prevent or treat delayed graft function. This study is designed to evaluate the safety and activity of an investigational drug in improving renal function in patients who have undergone renal transplantation and have signs and symptoms of significant renal injury and are at risk for dialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years of age
2. Had renal transplantation due to end stage disease requiring chronic dialysis
3. Study drug can be administered within 36 hours after transplantation
4. Received kidney from healthy donor or donor with history of diabetes mellitus or hypertension
5. Donor terminal serum creatinine ≤ 2.2 mg/dL.
6. No urine output, OR average urine output of < 50 cc/H over 8 or more consecutive hours, OR normal urine output following transplantation that diminished to average of < 50 cc/H over 8 or more consecutive hours, OR creatinine reduction ratio at 24 hours after transplantation to pre-transplantation is < 30%.
7. Reason for low urine output is unlikely due to structural changes. If clinically indicated, an ultrasound will be performed
8. Dry weight to< 120kg and BMI <35
9. Women of child bearing potential have a negative serum pregnancy test prior to transplantation.
10. Women of child bearing potential (including perimenopausal women who have had a menstrual period within 1 year) must agree to use 2 forms of effective birth control regimen (at least one-barrier method) during the 28-day study period. Men must agree to use condoms during the 28-day study period.
11. In the opinion of the investigator, the subject is capable of understanding and complying with the protocol.
12. Subjects must have signed the informed consent document prior to performance of any study related procedure including screening procedure.

Exclusion Criteria:

1. Subject with normal urine output and not requiring dialysis prior to renal transplantation (i.e., had pre-emptive renal transplantation).
2. Signs and symptoms of volume depletion.
3. Recipient of multiple organ transplantation or scheduled for multiple organ transplantation.
4. Recipient of pediatric en-bloc kidney transplantation.
5. Recipient of kidney with cold ischemia time > 40 hours
6. Has measurable donor-specific antibody or positive cross-match requiring deviation from standard immunosuppressive therapy.
7. Currently participating in or has participated in an investigational drug or medical device study within 30 days or five half-lives, whichever is longer, prior to enrollment into this study.
8. Concurrent sepsis or active bacterial infection.
9. Have an active malignancy or history of solid, metastatic or hematologic malignancy with the exception of basal or squamous cell carcinoma of the skin that has been removed.
10. Women of child bearing potential who are breast feeding.
11. History of positive HIV test.
12. History of rheumatoid arthritis.
13. Subjects who require the cytochrome P450 1A2 (CYP1A2) inhibitors, ciprofloxacin and/or fluvoxamine (Luvox®)
14. Subject is unwilling or unable to comply with the protocol or to cooperate fully with the Investigator or the site personnel.
15. Subject is not deemed medically stable for the study in the opinion of the Investigator or the subject's primary nephrologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-02; Primary Completion 2015-01 (Actual); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Urine production | 28 days
  mean time (days) until production of ≥ 50 cc/H of urine over a 12 hour period

SECONDARY OUTCOMES:
Change from baseline urine production | 28 days
  Change from baseline urine production (cc/H) at each of the following time points: Day 3, Day 7, Day 14, and Day 28
creatinine clearance | 28 days
  Mean measured 24-hour creatinine clearance at Days 3, 7, 14, and 28
Incidence of delayed graft function | 7 days
  Incidence of delayed graft function (required dialysis due to inadequate renal function during the 7 days after transplantation)
Number of dialysis sessions | 28 days
  Number of dialysis sessions through Day 7, 14, and 28
Daily urine output | 14 days
  Mean total daily urine output through Day 14
Mean serum creatinine | 28 days
  Mean serum creatinine at Days 4, 7, 10, 14, and 28
Number of acute rejection episodes | 28 days
  Number of acute rejection episodes
Length of hospitalization following transplantation | 28 days
  Length of hospitalization following transplantation
Biomarkers | 28 days
  Comparison of biomarkers
adverse events, clinical laboratory evaluations, vital signs, ECG results | 28 days
  Safety assessments include adverse events, clinical laboratory evaluations, vital signs, ECG results.

CONTACTS AND LOCATIONS:
Overall Officials: Weizhong Cai, PhD, Study Director — Sponsor GmbH
Locations (6):
- United States (6):
  - California Institute of Renal Research, San Diego, California
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Division of Transplant Surgery, University of Maryland School of Medicine, University of Maryland Medical Center, Baltimore, Maryland
  - State University of New York at Buffalo, Buffalo, New York
  - The Methodist Hospital, Houston, Texas